CLINICAL TRIAL: NCT02229110
Title: Effectiveness of a Computerised Prompt for Primary and Secondary Care Physicians to Refer or Refer Back Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Prof. G.E.H.M. Rutten, Professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-039/C
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus
Keywords: type 2 diabetes mellitus; e-Health; allocation of care; clinical inertia; quality of care; patient satisfaction
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Signal (Active Comparator): In addition to usual care, there will be an automatic signal in the electronic medical record (EMR) upon opening that will show the reader that the patient is currently not treated in the correct treatment setting and it simultaneously will give advice to which treatment allocation this patient should be transferred to.
  Interventions: Other: Signal
- No signal (No Intervention): Patients receive usual care, consisting of 4 office visits yearly

INTERVENTIONS:
Other: Signal — Automatic signal in the electronic medical record
  Arms: Signal

SUMMARY:
Patients with type 2 diabetes mellitus can receive care in the general practice or at the outpatient clinic. In the region of Amersfoort in The Netherlands, primary care practices and the hospital are connected through Diamuraal to organize the diabetes care in that region. They work in the same electronic medical record, and patients can request access to their own record (called a patient web portal). They set up Diamuraal guidelines, based on the guidelines of the Dutch College of General Practitioners and Internists, on where the patient care needs to be allocated (primary or secondary care), depending on the amount of specific care a patient needs. Despite guidelines, not all patients are treated in the correct place.

Our hypotheses is that when we improve triage we can cause a major shift from treatment in secondary care to primary care and from primary care to self-care by using the patient web portal. Furthermore, patients who needs extra attention due to problems with their diabetes or complications can receive this extra attention due to increased e-consultation between primary care and secondary care and if necessary actually can, during a short time, be treated by an internist. We hope to achieve this by introducing a signal in the electronic medical record. This signal allocates patients according to the guidelines and warns a physician if their patients is not treated according to that guideline. The health care provider can then discuss this situation with his patient. We believe that this leads to shift in allocation of care, in which optimal care is provided and patients are made more aware of their situation which hopefully leads to better self-management and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes mellitus
* health care provider work within Diamuraal setting

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2779 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The number of participants with change in allocation of care after intervention | One year
  One of the following:
  1. shift from primary care to secondary care
  2. shift from secondary care to primary care
  3. continuation of treatment in primary care but with addition of e-consultation with secondary care
  4. continuation of treatment in primary care but with replacement of one or more office visits in self-control

SECONDARY OUTCOMES:
Assembly of reasons by health care providers for not following the guidelines | One year
Change in quality of diabetes care | One year
  Measured with Quality of Care and Outcomes in Type 2 Diabetes scoring system (QuED) containing scores for biomedical data (HbA1c, blood pressure, lipids, medication regimen, number of measurements)
Change in diabetes treatment satisfaction | One year
  Measured with the diabetes treatment satisfaction questionnaire (DTSQ): six questions on satisfaction with treatment regimen and two questions on perceived frequency of hyperglycemia and hypoglycemia.
Number of participants who meet their treatment goals | One year
  Measured in number of goals that are met

CONTACTS AND LOCATIONS:
Overall Officials: Guy EH Rutten, MD PhD, Principal Investigator — UMC Utrecht; Lioe-Ting Dijkhorst-Oei, MD, PhD, Study Director — UMC Utrecht; Maaike CM Ronda, MD, Study Director — UMC Utrecht
Locations (2):
- Netherlands (2):
  - Diamuraal-associated GP practices, Amersfoort
  - Meander Medical Center, Amersfoort

REFERENCES:
- [Background] Ronda MC, Dijkhorst-Oei LT, Gorter KJ, Beulens JW, Rutten GE. Differences between diabetes patients who are interested or not in the use of a patient Web portal. Diabetes Technol Ther. 2013 Jul;15(7):556-63. doi: 10.1089/dia.2013.0023. Epub 2013 Jun 18. PMID 23777369
- See also: Related Info — http://www.diamuraal.nl